CLINICAL TRIAL: NCT05823415
Title: Clinical Evaluation of Laterally Closed Tunnel Technique Versus Coronally Advanced Flap Combined With Connective Tissue Graft for the Treatment of Isolated RT2 Gingival Recession: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Laterally Closed Tunnel Technique Versus Coronally Advanced Flap Combined With Connective Tissue Graft for the Treatment of Isolated RT2 Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sarah Rajab, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241953
Record Dates: First submitted 2023-02-16; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laterally closed tunnel technique with CTG (Experimental)
  Interventions: Procedure: Laterally Closed Tunnel with CTG
- Coronally advanced flap with CTG (Active Comparator)
  Interventions: Procedure: CAF with CTG

INTERVENTIONS:
Procedure: Laterally Closed Tunnel with CTG — A novel minimally invasive surgical approach laterally closed tunnel technique (LCT) has been recently introduced for the management of isolated gingival recession. The laterally closed tunnel technique ensures predictability by tunneling and mobilization of flap for graft coverage.
  Arms: Laterally closed tunnel technique with CTG
Procedure: CAF with CTG — Gold standard surgical technique
  Arms: Coronally advanced flap with CTG

SUMMARY:
The aim of this study is to evaluate reduction of recession depth using lateral closed tunnel technique versus CAF technique using connective tissue graft in single RT2 gingival recession cases.

ELIGIBILITY:
Inclusion Criteria:

* Single RT2 buccal gingival recession ≥ 2 mm in the esthetic zone (Gingival recession associated with loss of inter-proximal attachment. The amount of interproximal attachment loss (measured from the interproximal CEJ to the depth of the interproximal pocket) was less than or equal to the buccal attachment loss (measured from the buccal CEJ to the depth of the buccal pocket)
* Patients with good oral hygiene
* Medically free patients
* No signs of active periodontal disease (with no site showing probing depth > 4 mm and full-mouth bleeding score (FMBS) 20% (measured at four sites per tooth).
* Palate with sufficient thickness to accommodate soft tissue defect.

Exclusion Criteria:

* Smokers
* Pregnancy
* Severe gag reflex
* Non-carious cervical lesion
* History of mucogingival or periodontal surgery at the experimental site
* History of medication that can affect periodontal healing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in recession depth | 6 Months

SECONDARY OUTCOMES:
Post-operative pain assessed by VAS Scale | 2 week
  Pain score reported by the patient directly through Visual Analogue Scale score (between 0 and 10, 0: no pain, 1: minimal pain 5: moderate pain, 10: severe pain)
Probing Depth | 6 months
Clinical Attachment Level | 6 months
  will be measured by a periodontal probe
Width of Keratinized Tissue | 6 months
Gingival Thickness | 6 months
Percentage of complete root coverage by williams periodontal probe | 6 months
  Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100

IPD SHARING:
Plan to Share IPD: Undecided